CLINICAL TRIAL: NCT05598216
Title: LDL Cholesterol: Friedewald, Always the Best Option to Evaluate LDL cholesteRol Concentration in norMal and Dyslipidemic sUbjects, in Fasting and Pot-prandiaL State?
Brief Title: Assessment of Different Equations to Accurately Calculate LDL Cholesterol
Acronym: LDL FORMULA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 488
Record Dates: First submitted 2022-10-17; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Dyslipidemias; Lipid Disorder
Keywords: LDL cholesterol; equation; postprandial; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fasting state: based on the sampling time and the serum's aspect
  Interventions: Diagnostic Test: no intervention, Serum LDL cholesterol calculation
- non-fasting state: based on the sampling time and the serum's aspect
  Interventions: Diagnostic Test: no intervention, Serum LDL cholesterol calculation

INTERVENTIONS:
Diagnostic Test: no intervention, Serum LDL cholesterol calculation — The serum LDL cholesterol concentrations will be calculated using at least three different equations (Friedewald, Sampson, Martin-Hopkins)

SUMMARY:
Purpose The LDL-C is a very important marker of the lipid panel which allows the introduction of a treatment and then the follow-up to prevent the cardiovascular risk. Friedewald et al have established the most widely used equation at the present time. However, it has many well-known limitations, as being false in postprandial period.

New equations have been developed recently. Our work consisted in the assessment of the accuracy of Friedewald, Sampson and Martin-Hopkins equations and evaluated the consequences in terms of misclassification. Given that European recommendations allow the realization of lipid profiles in postprandial period, we studied the accuracy of these equations in non-fasting state .

Method The LDL cholesterol concentrations will be calculated using at least three different equations (Friedewald, Sampson, Martin-Hopkins). Results will be compared between equations and between calculated and measured concentrations determined using an ultracentrifugation method. The study is conducted out according to The Code of Ethics of the World Medical Association (Declaration of Helsinki) and obtained the agreement of the Scientific and Ethics Committee of the Hospices Civils de Lyon (LDL EQUATION CNIL 21_488) Hypothesis

To evaluate the most accurate equation in different conditions:

* Fasting and non-fasting state
* In subjects with normal or dyslipidemic lipid profile To evaluate the clinical impact on risk re-classification and lipid treatment goals if LDL-c is calculated using the best equation instead of the Friedewald's.

ELIGIBILITY:
Inclusion Criteria:

* lipid profile performed in the location 1 during the recruitment period

Exclusion Criteria:

* Results outside the first and 99th percentile for TG parameters
* Samples slightly opalescent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: lipid profile performed in the lab during the recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 160000 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the most accurate equation to calculate LDL cholesterol (mmo/L or g/L) | The outcome measure will be assessed through study completion, an average of 1 year
  The outcome measure is LDL cholesterol concentration (mmol/l or g/L) determined using different equations (Friedwald, Martin Hopkins, Sampson equations, …) and measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire de Biologie Médicale Multi Sites, Centre de Biologie et de Pathologie Est, Bron, France

REFERENCES:
- [Derived] Vasse J, Lassartesse A, Marmontel O, Charriere S, Bouveyron C, Marrie N, Moulin P, Di Filippo M. Assessment of three equations to calculate plasma LDL cholesterol concentration in fasting and non-fasting hypertriglyceridemic patients. Clin Chem Lab Med. 2023 Sep 8;62(2):270-279. doi: 10.1515/cclm-2023-0360. Print 2024 Jan 26. PMID 37678263